CLINICAL TRIAL: NCT00213421
Title: Comparison of Two Therapeutic Strategies of Dermoval in Treatment of Bullous Pemphigus
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2000/014/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
  Interventions: Drug: Dermoval
- 2
  Interventions: Drug: Dermoval

INTERVENTIONS:
Drug: Dermoval — group 1 elevated corticosteroids : attack treatment 2 tubes of 10g (4t/d) decreasing treatment : one month: 2 tubes/J (2t/d); 2 months : 2 tubes 1d sur 2 (1d/j); 4 months : 2 tubes 2 fois /week (0,6t/d); 4 months : 2 tubes 1 fois /week (0,3t/d)fois /week (0,3t/d) group 2 low corticosteroids : for paucibullous form with weight < 45kg attack treatment 1 tubes of 10g (1t/d)decreasing treatment 1 month : 1 tube every 2d (0,5t/d; 1 month : 1 tubes 2 fois /week (0,3t/d) 1 month : 1 tubes 1 fois/week (0,15t/d); for paucibullous form with weight > 45kg or for multibullous form with weight < 45kg attack treatment 2 tubes of 10g (2t/d)decreasing treatment 1 month : 2 tubes every 2j (1t/d; 1 month : 2 tubes 2 fois /week (0,6t/d) 1 month : 2 tubes 1 fois /week (0,3t/d)and for multibullous form attack with weigth > 45kg treatment 3 tubes of 10g (3t/d)decreasing treatment 1 month : 3 tubes every 2days (1,5t/d) 1 month : 3 tubes 2 fois /week (1t/j)1 mois : 3 tubes 1 fois /week (0,45t/d)

SUMMARY:
to compare efficacity and tolerance of two stratégies of dermoval application in treatment of bullous pemphigus.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* immunoflurescence, histological exam, predictive value according to bullous pemphigus diagnostic
* consentment patient

Exclusion Criteria:

* age < 18
* no consentment
* localized bullous pemphigus (<400cm2)
* linear IgA pemphigus
* corticothérapy, immunotherapy
* pregnant woman pemphigus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with compatible bullous pemphigoid clinical exam
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2001-08; Primary Completion 2004-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Joly, MD-PHD, Principal Investigator — UH Rouen
Locations (1):
- UH-rouen, Rouen, Seine maritime, France